CLINICAL TRIAL: NCT01476592
Title: A Biological Study of Resveratrol's Effects on Notch-1 Signaling in Subjects With Low Grade Gastrointestinal Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0097; OS10325 (Other: University of Wisconsin Carbone Cancer Center); 2011-0097 (Other: Institutional Review Board); A539740 (Other: UW Madison); SMPH\SURGERY\GEN SURG (Other: UW Madison); NCI-2011-03685 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2011-11-09; First posted 2011-11-22 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2018-11

CONDITIONS: Neuroendocrine Tumor
Keywords: gastrointestinal neuroendocrine tumor
MeSH Terms: conditions — Neuroendocrine Tumors; Gastro-enteropancreatic neuroendocrine tumor | interventions — Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resveratrol (Experimental): 5 gm/day of resveratrol orally, in two divided doses of 2.5 gm each without a break in therapy for a total of three cycles.
  Interventions: Dietary Supplement: Resveratrol

INTERVENTIONS:
Dietary Supplement: Resveratrol — 5 gm/day of resveratrol orally, in two divided doses of 2.5 gm each without a break in therapy for a total of three cycles.

SUMMARY:
Resveratrol has been shown to activate a protein called Notch-1. Signaling of Notch-1 has been shown to prevent tumor cell growth. Resveratrol has also been shown to prevent growth of tumors in mice. The purpose of this study is to examine the effects of resveratrol and Notch-1 on neuroendocrine tumor tissue and to examine how people with neuroendocrine tumors who take resveratrol for up to three months tolerate the product.

DETAILED DESCRIPTION:
Patients will be treated with a dose of 5 gm/day of resveratrol orally, in two divided doses of 2.5 gm each without a break in therapy for a total of three cycles. All patients who receive at least one dose of resveratrol will be evaluated for toxicity and tolerability. Toxicities will be assessed every 28 days while the study drug is being taken by the patient. Pill bottles will be reviewed at this visit as well to ensure compliance with the study medication. Toxicities will be graded according to the NCI Common Toxicity Criteria. Blood will be drawn for a complete blood count and comprehensive metabolic panel. In addition, one vial of serum will be stored at the time of each toxicity assessment for later analysis of resveratrol levels. This level must be drawn one hour after the morning dose and the participants will be instructed to alter the time of the morning dose so as to allow proper timing with the scheduled blood draw.

During the third cycle of treatment, a post-treatment biopsy will be obtained for study related purposes and will be processed only for research related purposes.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status of 0-2
2. Age >18 years old
3. Women who are not postmenopausal must have a negative enrollment blood test and agree to use an effective mode of contraception while taking the study medication
4. Greater than four weeks must have elapsed since any previous therapy was administered for the neuroendocrine tumor, including surgery, radiation, chemotherapy or local liver therapy.
5. Octreotide use is allowed but must be initiated at least four weeks prior to enrollment and to the pre-treatment biopsy
6. Able to give informed consent and willing to undergo the post-treatment research biopsy
7. Must be able to take oral medications and be without GI tract obstructive symptoms
8. Subjects with another malignancy for which they are either undergoing treatment with chemotherapy or radiation, or with a malignancy for which such treatments have been recommended, would be excluded or withdrawn from the study.
9. Must agree to abstain from excessive alcohol, as defined by greater than the equivalent of three glasses of wine per day or one six pack of beer per day

Exclusion Criteria:

1. The principal investigator will review each subject's current medications prior to enrollment of the study to ensure that the administration of Resveratrol will not affect their current medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Notch1 activation in post-treatment tumor biopsy specimens when compared to pretreatment levels | 1 year
  1. The investigators aim primarily to show that resveratrol therapy in patients with low-grade GI neuroendocrine tumors will significantly increase Notch1 activation in post-treatment tumor biopsy specimens when compared to pretreatment levels.
  Endpoints: The primary endpoint will be the level of expression of full length Notch1, cleaved Notch1, HES-1, and ASCL-1, as measured by Western blot using quantitative densitometry. The pre-treatment and post-treatment biopsies will be processed and analyzed simultaneously so as to minimize inter-test variability.

SECONDARY OUTCOMES:
Demonstrate that resveratrol at 5 gm per day will be well tolerated with minimal dose limiting toxicities in this patient population. | 1 year
  Frequency of grade three or greater toxicities as defined by the NCI Common Toxicity Criteria.
Describe the effect of resveratrol on tumor growth as demonstrated by standard cross sectional imaging and tumor markers. | 1 year
  The level of tumor markers (eg, chromogranin, 5-HIAA, gastrin, and others) pre-treatment will be compared to the post-treatment levels (collected every three months) as a measure of tumor response. In addition, serial axial imaging will be used to document tumor response rates according to standard Response Evaluation Criteria in Solid Tumors (RECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Emily R. Winslow, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/